CLINICAL TRIAL: NCT00541086
Title: A Phase III Study Comparing Anastrozole, Letrozole and Exemestane, Upfront (for 5 Years) or Sequentially (for 3 Years After 2 Years of Tamoxifen), as Adjuvant Treatment of Postmenopausal Patients With Endocrine-responsive Breast Cancer
Brief Title: Study of Anastrozole, Letrozole, or Exemestane With or Without Tamoxifen in Treating Postmenopausal Women With Hormone-Responsive Breast Cancer That Has Been Completely Removed By Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Gruppo Italiano Mammella (GIM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000570041; GIM-3-FATA; EUDRACT-2006-004018-42; EU-20764
Record Dates: First submitted 2007-10-05; First posted 2007-10-08 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; estrogen receptor-positive breast cancer; progesterone receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; exemestane; Letrozole; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- A - anastrozole (Experimental): Up-front adjuvant anastrozole for 5 years
  Interventions: Drug: anastrozole
- B - exemestane (Experimental): Up-front adjuvant exemestane for 5 years
  Interventions: Drug: exemestane
- C - letrozole (Experimental): Up-front adjuvant letrozole for 5 years
  Interventions: Drug: letrozole
- D - tamoxifen followed by anastrozole (Active Comparator): Switch adjuvant treatment with tamoxifen for 2 years followed by anastrozole for 3 years
  Interventions: Drug: anastrozole; Drug: tamoxifen citrate
- E - tamoxifen followed by exemestane (Active Comparator): Switch adjuvant treatment with tamoxifen for 2 years followed by exemestane for 3 years
  Interventions: Drug: exemestane; Drug: tamoxifen citrate
- F - tamoxifen followed by letrozole (Active Comparator): Switch adjuvant treatment with tamoxifen for 2 years followed by letrozolefor 3 years
  Interventions: Drug: letrozole; Drug: tamoxifen citrate

INTERVENTIONS:
Drug: anastrozole — 1 mg per day, orally
  Arms: A - anastrozole; D - tamoxifen followed by anastrozole
Drug: exemestane — 25 mg per day, orally
  Arms: B - exemestane; E - tamoxifen followed by exemestane
Drug: letrozole — 2.5 mg per day, orally
  Arms: C - letrozole; F - tamoxifen followed by letrozole
Drug: tamoxifen citrate — 20 mg per day, orally
  Arms: D - tamoxifen followed by anastrozole; E - tamoxifen followed by exemestane; F - tamoxifen followed by letrozole

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking use of estrogen by the tumor cells. Anastrozole, letrozole, and exemestane may fight breast cancer by lowering the amount of estrogen the body makes. It is not yet known whether giving tamoxifen followed by anastrozole, letrozole, or exemestane is more effective than giving anastrozole, letrozole, or exemestane alone in treating breast cancer.

PURPOSE: This randomized phase III trial is studying giving tamoxifen followed by either anastrozole, letrozole, or exemestane to see how well it works compared to anastrozole, letrozole, or exemestane alone in treating postmenopausal women with hormone-responsive invasive breast cancer that has been completely removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare sequential tamoxifen for 2 years followed by anastrozole, letrozole, or exemestane for 3 years vs anastrozole, letrozole, or exemestane for 5 years in terms of disease-free survival in postmenopausal women with nonrecurrent, nonmetastatic invasive endocrine-responsive breast cancer.
* To compare disease-free survival in patients treated with anastrozole vs letrozole vs exemestane.

OUTLINE: This is a multicenter study. Patients are stratified according to hormone receptor status (estrogen receptor [ER]-positive and progesterone [PgR] receptor-positive disease vs ER-positive and PgR-negative disease vs ER-negative and PgR-positive disease vs ER- or PgR-positive disease or ER or PgR status unknown), HER-2/neu status (positive [3+ by IHC or positive by fluorescence in situ hybridization ( FISH)] vs negative vs unknown), prior chemotherapy (none vs adjuvant vs neoadjuvant vs both adjuvant and neoadjuvant), and nodal status (pN0 vs pN1 vs pN2 vs pN3). Patients are randomized to 1 of 6 treatment arms.

* Arm I: Patients receive oral anastrozole once daily for 5 years.
* Arm II: Patients receive oral exemestane once daily for 5 years.
* Arm III: Patients receive oral letrozole once daily for 5 years.
* Arm IV: Patients receive oral tamoxifen citrate once daily for 2 years followed by oral anastrazole once daily for 3 years.
* Arm V: Patients receive oral tamoxifen citrate once daily for 2 years followed by oral exemestane once daily for 3 years.
* Arm VI: Patients receive oral tamoxifen citrate once daily for 2 years followed by oral letrozole once daily for 3 years.

Treatment in all arms continues in the absence of disease recurrence or unacceptable toxicity.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast cancer completely removed by surgery

  * Any T, any N
  * No recurrent or metastatic disease
* Estrogen or progesterone receptor-positive disease in primary tumor, as defined by 1 of the following:

  * At least 10% of tumor cells positive by immunohistochemistry
  * At least 10 fmol/mg cytosol protein by ligand binding assay
* Patients with HER-2/neu positive tumors are eligible provided they receive trastuzumab (Herceptin®) according to the registered schedule

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal, defined by ≥ 1 of the following:

  * Age ≥ 60 years
  * Age 45-59 and satisfying 1 or more of the following criteria:

    * Amenorrhea for ≥ 12 months AND intact uterus
    * Amenorrhea (secondary to hysterectomy, hormone replacement therapy (HRT), or chemotherapy) for < 12 months AND follicle-stimulating hormone within the postmenopausal range
  * Underwent prior bilateral oophorectomy at any age >18 years
* No concurrent illness that contraindicates adjuvant endocrine treatment
* No other invasive breast cancer or invasive malignancy within the past 10 years, except adequately cone-biopsied squamous cell or basal cell skin cancer or carcinoma in situ of the cervix
* No concurrent disease that would place the patient at unusual risk

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Adjuvant or neoadjuvant chemotherapy must be completed prior to study entry
* At least 1 month since prior and no concurrent HRT
* More than 30 days since prior systemic investigational drugs
* No prior tamoxifen as part of any breast cancer prevention study
* Prior or concurrent locoregional radiotherapy allowed
* No other concurrent experimental drugs
* No concurrent bisphosphonates, unless indicated as treatment for osteoporosis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3697 (Actual)
Dates: Start 2007-03 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years

SECONDARY OUTCOMES:
Overall Survival | 5 years
Distant metastasis-free survival | 5 years
Cumulative incidence of contralateral breast cancer as first event | 5 years
Breast cancer-free survival | 5 years
Cumulative incidence and type of second non-breast invasive cancer | 5 years
Effects on lipid profile | 5 years
Toxicity as assessed by NCI CTCAE v3.0 | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Sabino De Placido, MD, Study Chair — Federico II University
Locations (5):
- Italy (5):
  - Federico II University Medical School, Naples
  - Istituto Nazionale per lo Studio e la Cura dei Tumori, Naples
  - Seconda Universita di Napoli, Naples
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Istituti Fisioterapici Ospitalieri - Roma, Rome

REFERENCES:
- [Derived] De Placido S, Gallo C, De Laurentiis M, Bisagni G, Arpino G, Sarobba MG, Riccardi F, Russo A, Del Mastro L, Cogoni AA, Cognetti F, Gori S, Foglietta J, Frassoldati A, Amoroso D, Laudadio L, Moscetti L, Montemurro F, Verusio C, Bernardo A, Lorusso V, Gravina A, Moretti G, Lauria R, Lai A, Mocerino C, Rizzo S, Nuzzo F, Carlini P, Perrone F; GIM Investigators. Adjuvant anastrozole versus exemestane versus letrozole, upfront or after 2 years of tamoxifen, in endocrine-sensitive breast cancer (FATA-GIM3): a randomised, phase 3 trial. Lancet Oncol. 2018 Apr;19(4):474-485. doi: 10.1016/S1470-2045(18)30116-5. Epub 2018 Feb 23. PMID 29482983